CLINICAL TRIAL: NCT04562103
Title: Comparison of Ropivacaine Plasma Concentration With or Without Epinephrine for Posterior Quadratus Lumborum Block in Cesarean Section
Brief Title: Ropivacaine Plasma Concentration With or Without Epinephrine for Posterior Quadratus Lumborum Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ID 2979
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-07

CONDITIONS: Local Anesthetic Systemic Toxicity; Anesthesia, Local
Keywords: Quadratus lomborum block; Ropivacaine; Epinephrine
MeSH Terms: interventions — Epinephrine; Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epinephrine QLB (Experimental): In this group quadratus lomborum block was performed with 0.375% ropivacaine+100 mcg epinephrine.
  Interventions: Drug: Epinephrine / Ropivacaine
- Plane QLB (Active Comparator): In this group quadratus lomborum block was performed with plane 0.375% ropivacaine.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Epinephrine / Ropivacaine — In this group quadratus lomborum block was performed with 0.375% ropivacaine+100 mcg epinephrine.
  Arms: Epinephrine QLB
Drug: Ropivacaine — In this group quadratus lomborum block was performed with plane 0.375% ropivacaine.
  Arms: Plane QLB

SUMMARY:
Introduction The posterior Quadratus Lumborum Block (pQLB) has been used in postoperative pain management after Cesarean Section (CS). However, there are no data about pQLB safety in pregnants, at increased risk of local anesthetic systemic toxicity (LAST). The purpose of the present study was to explore the efficacy and the safety of adding epinephrine to ropivacaine for bilateral pQLB vs. bilateral pQLB performed with ropivacaine alone in CS.

Methods Fifty-two pregnants were consecutively allocated to one of 2 groups [e-pQLB (0.375% ropivacaine+100 mcg epinephrine) or pQLB (0.375% ropivacaine)] and the investigators evaluated if the adjunct of epinephrine to ropivacaine increases of efficacy (measured as opioid consumption during the first 24 postoperative hours, time for first request of opioid and pain values reported by patients) and the safety (measured as peak and plasmatic concentration of ropivacaine) of pQLB.

DETAILED DESCRIPTION:
BACKGROUND The posterior Quadratus Lumborum Block (pQLB) is a posterior abdominal wall block in which local anesthetic (LA), administered posteriorly to Quadratus Lumborum (QL) muscle, spreads underneath intermedium layer of thoracolumbar fascia, into a triangular space named lumbar interfacial triangle. This interfascial plane is in close relation to thoracic paravertebral (PV) space. Local anesthetic spread into this space could explain analgesic efficacy of pQLB1. Compared to lateral QLB, in which LA is administered laterally to QL muscle, pQLB is safer (needle tip is separated from the peritoneum by QL muscle) and easier to perform (injection point is more superficial). Posterior QLB efficacy has been demonstrated in major abdominal surgery. In Cesarean Section (CS) pQLB efficacy vs placebo and superior efficacy vs TAP block was showed. Ropivacaine arterial concentration after QLB, in laparoscopic gynaecological surgery has been studied. To the best of our knowledge no author investigated pQLB safety in obstetric population, at increased risk of local anesthetic systemic toxicity (LAST) because of physiological modifications occurring during pregnancy (increased cardiac output, increased arterial and venous blood tissue flow, decreased concentration of plasma binding protein). Adding epinephrine to local anesthetic, determining a delayed AL systemic reabsorption and a reduced plasmatic concentration, could improve pQLB efficacy and safety, as demonstrated for Transversus Abdominal Plain (TAP) block and sciatic and femoral block.

METHODS Patients were consecutively allocated into one of two groups: e-pQLB (0.375% ropivacaine+ 100 mcg epinephrine) or pQLB (0.375% ropivacaine). Before surgery, under local anesthesia, 2 venous accesses were founded, one for fluids and drugs injection and the second one, contralaterally, for venous samples only. During surgical procedure standard hemodynamic monitoring was provided; fetal wellbeing was registered by cardiotocographic monitoring. Supplemental oxygen has was provided by Venturi mask. SA was administered in sitting position, at L3-4 lumbar interspace, using hyperbaric bupivacaine 0.5% 9 mg plus sufentanil 5 mcg. Surgical procedure started when T4 level has been reached. Posterior QLB was administered at the end of surgical procedure, with patient in supine position, under monitoring and after cleaning the skin with surgical solution (ChloraPrep, Carefusion, 244 LTD, UK). A Sonosite M-Turbo echograph ( FUJIFILM Sonosite Europe, Amsterdam, Netherlands) and a broadband (5-8 MHz) convex probe covered with a sterile plastic sheath have been used. The probe was placed at the level of the anterior superior iliac spine and moved cranially until the three abdominal wall muscles were identified. The external oblique muscle was followed posterolaterally until its posterior border was found. The probe was tilted down to identify the bright hyperechoic line that corresponds with the intermediate layer of the thoracolumbar fascia. The needle (Ultraplex 360, B.Braun Melsungen, Germany) was inserted in plane from medial (anterior) to lateral (posterior). The optimal point of injection was determined using hydrodissection. In e-pQLB group ropivacaine 0.375%+epinephrine 100 mcg 20 ml for each side was administered; in pQLB group ropivacaine 0.375% 20 ml for each side was administered. After block, venous samples (2 ml each) were performed at 10, 30, 45, 60, 120 minutes. The ropivacaine concentration was set at 2.2 mcg/ml, which represents the venous threshold value of systemic toxicity14. To evaluate LAST patients have been asked for perioral tingling, metallic taste, tinnitus, visual disturbance or slurred speech at the time that each blood sample has been obtained.

Intraoperative ketorolac 30 mg and acetaminophen 1 g were administered. After surgery, in Post Anesthesia Care Unit (PACU), a PCA pump was connected to patients and programmed to deliver 1 mg morphine bolus on demand with a lock out interval of 8 min and no background infusion. All patients received regular intravenous paracetamol 1g 6 hourly and intravenous ketorolac 30 mg 12 hourly.

Experimental procedure Chemicals, reagents and equipment Methanol and acetonitrile were HPLC grade and were purchased from VWR Chemicals (Radnor, PA, USA). Water was purified by Millipore Synergy-UV-System (Bedford, MA, USA). 20 % ammonium hydroxide solution was provided by Carlo Erba Reagents (Milan, Italy), acetic acid 99-100% and phosphoric acid ≥ 85% were provided by Sigma-Aldrich (St. Louis, MO, USA). Ropivacaine and Ropivacaine-d7 hydrochloride (used as internal standard, IS) were purchased by USP (Rockville, MD, USA) and Toronto Research Chemicals (North York, ON, Canada), respectively. Neostigmine methylsulphate was provided by LGC Standards (Luckenwalde, Germany).OASIS HLB SPE cartridges (3 mL, 60 mg) were supplied by Waters (Milford, MA, USA). PTFE disposable filters (0.45 µm) were purchased from Membrane solutions (Plano, TX, USA). Visiprep DL SPE Vacuum Manifold was purchased by Supelco/Sigma-Aldrich (St. Louis, MO, USA). The heating block "Pierce - Reacti-Therm III" was purchased from ThermoFisher Scientific (Waltham, MA, USA). Centrifuge 5415D supplied by Eppendorf (Hamburg, Germany).1 mg mL-1 stock solutions of ropivacaine and ropivacaine-d7 were prepared in methanol. Working standard solution dilutions were prepared from these latter solutions and were finally diluted by serial dilution to spike blank plasma samples for the construction of matrix-matched calibration curve in order to have final ropivacaine concentrations in the interval of 0.8 - 13.2 ng mL-1. Working solutions were stored at -20 °C and prepared daily. Stock solutions were analysed regularly up to six month after the preparation to assess their stability in the time and whether there was degradation of the analytes.

Plasma sampling Patients' blood samples (5 mL) were collected in tubes containing ethylenediaminetetraacetic acid (EDTA) and were added to 25 µL of 20 mg mL-1 neostigmine methylsulfate solution to block esterase activity in the plasma14. The samples were stored in ice-water bath for 10-15 min and then centrifuged at 1300 × g at 4°C for 5 min to obtain plasma. Collected plasma samples were stored at -20 °C until analyzed.

Sample preparation A modified procedure of Toonoka K was used. A 0.2-mL-aliquot of plasma sample was added to 0.3 mL of purified water and vortex-mixed. The diluted sample was spiked with 25 µL of a methanolic solution of ropivacaine-d7 (IS) (85.0 ng mL-1) and added to 0.5 mL of 4 % phosphoric acid solution. The mixture was vortex-mixed and centrifuged (16110 × g, 2 min). The supernatant is then loaded on the OASIS HLB SPE cartridge which was previously conditioned with 2 mL of methanol and equilibrated with 2 mL of purified water. After the washing steps with 2 mL of 5% methanol solution and 2 mL of 2% ammonium hydroxide in a 10% methanol solution, sample was eluted with 2 mL of methanol/ 2% acetic acid (70/30, v/v) solution. The extract was next evaporated under a stream of nitrogen at 30°C and the dry residue was dissolved in 0.2 mL of the mobile phase and filtrated prior to LC-MS/MS analysis (10 μL injection).

LC-MS/MS analysis Analyses were carried out using a LC system Perkin Elmer Series 200 Micro Pump equipped with a PE Series 200 auto sampler (Perkin Elmer, USA). The chromatographic separations were obtained under gradient conditions at room temperature (25°C) using a reverse phase HPLC column Kinetex 2.6 µm EVO C18 100 Å (100 × 3 mm) (Phenomenex, USA) with C18 guard column (4 mm × 2 mm) (Security Guard, Phenomenex, USA). The mobile phase was composed of ammonium hydroxide 0.53 mM pH 10.3 (mobile phase A) and acetonitrile (mobile phase B) and the flow rate was 0.3 mL min-1. The gradient profile began at 70 % A and held for 1 min, then changed to 25 % in 2 min and held for 3 min. The profile returned to 70 % A in 1 min and held for 1 min (total run: 8 min).

The API 3000 triple quadrupole mass spectrometer (AB Sciex, Canada) was equipped with an Electro Spray Ionization (ESI) source, and was set in positive ionization mode (source temperature: 450 °C; ionspray voltage: 5500 V; ultra-pure nitrogen as curtain and collision gas; ultra-pure air as nebulizer and auxiliary gas). One precursor ion and two product ions (two transitions) for ropivacaine and ropivacaine-d7 were monitored by MRM (Multiple Reaction Monitoring): 275.2 m/z > 126.1 m/z (most abundant ion used for quantification) and 275.2 m/z > 84.2 m/z (Figure 1). Collision energy (CE), declustering potential (DP), entrance potential (EP), and collision cell exit potential (CXP) were adjusted in MRM mode for each transition monitored in order to reach the highest sensitivity for all the analytes.

Plasma samples, used for the construction of five points matrix-matched calibration curves, were previously tested and shown to contain no residues of the compounds of interest. The ropivacaine concentration levels were set as follows: 0.82, 1.64, 3.28, 6.56 and 13.12 ng mL-1. The correlation between concentration and the detector response was determined by using a weighted (1/x) linear regression model (equation y = 0.117x + 0.00409; correlation coefficient r > 0.998; relative accuracy percentage for each point of the curve within the ± 5 % of the expected concentrations). Sample was appropriately further diluted to obtain concentrations of ropivacaine within the calibration ranges.

The main performance characteristics of the method were evaluated. Limit of detection (LOD) and limit of quantification (LOQ) values were 0.30 and 0.82 ng mL-1 of ropivacaine, respectively. Repeatability expressed as intra-day coefficient of variation (CV %) was in the interval of 1.99 - 11.44 % whereas intermediate precision expressed as inter-day CV % was in the interval 7.61 - 13.60 %. Recovery percentages were 99.03 - 110.7 %.

Statistical analysis Sample size estimation was based on a recent article from Hansen et al, who demonstrated that transmuscular quadratus lumborum block for elective CS significantly reduces postoperative opioid consumption and prolongs time to first opioid request when compared to placebo. In this single-center, randomized, placebo-controlled study, the mean 24 hours postoperative oral morphine equivalents was 65,3 mg vs 94,3 mg in the control group. Our primary hypothesis was that epinephrine added to ropivacaine for pQLB would result in a minimum 30% reduction of opioid consumption in the first 24 postoperative hours. Based on previous studies on opioid consumption, a SD of 40% was estimated. A sample size of at least 35 patients would give 80% power to detect a 30% reduction in opioid consumption, using t-tests with α=0,05. Fifty-two patients, twenty-six per group were included in the study to allow missing data or dropouts. The analysis was performed using Stata IC/15.1 (Stata Corp) and Microsoft Excel. Ordinal data and continuous data were analyzed using Wilcoxon rank sum test and Student's t-test as appropriate. Shapiro-Wilk test was used to assess normality of data distribution and the sd-test to verify equality of variances. For non-normally distributed data, a Mann-Whitney test was performed. Differences between categorical data were analyzed using the χ 2 or Fisher's exact test. Variables were presented as means (SD) or median (range). The data were given as ratio of means and 95% confidence intervals (CIs).A mixed-effects model for repeated measures ANOVA was used to assess the treatment-by time interaction; the p value included Box's conservative F test for the lack of compound symmetry assumption. The investigators applied log-rank tests to compare Kaplan-Meier plots, for duration of time until first analgesic request. Statistical significance level was 0.05%.

ELIGIBILITY:
Inclusion Criteria:

* first singleton pregnancy at term
* American Society of Anesthesiologists (ASA) physical status II;
* caesarean section under Spinal Anesthesia

Exclusion Criteria:

* patients enable to comprehend or use the verbal rating pain scoring system or patient controlled analgesia (PCA) pump;
* congenital coagulopathy;
* anatomical abnormalities;
* localized infections;
* use of drugs interfering with ropivacaine metabolism.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Caesarean Section
Enrollment: 52 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | at 6, 12 and 24 hours after the end of surgery
  To evaluate if the adjunct of epinephrine to local anesthetic would results in a reduction in postoperative pain compared to the block performed with ropivacaine alone. Pain at rest and with movement recorded with a visual analogue scale (from 0 to 10).
Postoperative analgesic requirement | First 24 hours after the end of surgery
  To evaluate if the adjunct of epinephrine to local anesthetic would results in a longer sensory block duration compared to the block performed with ropivacaine alone. Time between the block and first opioid analgesic requirement (minutes).

SECONDARY OUTCOMES:
Plasmatic concentration of Ropivacaine | At 10, 30, 45, 60, 120 minutes after the block
  To evaluate if adding epinephrine to local anesthetic reduces reabsorption and consequently the peak and the median venous plasmatic concentration of ropivacaine.
  Ropivacaine plasmatic concentration (mcg/ml) in the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico Agostino Gemelli, Rome, Italy